CLINICAL TRIAL: NCT02663804
Title: Total Knee Arthroplasty: Relation Between Patient Satisfaction and Implant Geometry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC/2014/0023
Record Dates: First submitted 2016-01-07; First posted 2016-01-26 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Osteoarthritis
Keywords: Total Knee Arthroplasty; Patient Satisfaction; PROMs; Implant Design
MeSH Terms: conditions — Osteoarthritis; Patient Satisfaction | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Care Provider

ARMS (3):
- Implant design 1 (Active Comparator): Journey II, BCS, Smith&Nephew
  Interventions: Device: Total Knee Arthroplasty
- Implant design 2 (Active Comparator): Persona, Zimmer
  Interventions: Device: Total Knee Arthroplasty
- Implant design 3 (Active Comparator): Unity, Corin
  Interventions: Device: Total Knee Arthroplasty

INTERVENTIONS:
Device: Total Knee Arthroplasty
  Other Names: Journey II, Smith&Nephew; Persona, Zimmer; Unity, Corin

SUMMARY:
A RCT (randomized controlled trial) comparing 3 different TKA (total knee arthroplasty) implant designs and investigating the relation between patient satisfaction and the implant geometry.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients of all ages, scheduled for TKA
* Primary osteoarthritis of the knee joint
* post traumatic arthritis
* rheumatoid arthritis

Exclusion Criteria:

* previous TKA in same joint
* evidence of neuromuscular or neurosensory deficiency
* immunologic suppression

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2014-04; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | Preop
  Determining patient specific factors by use of validated questionnaires
Patient Satisfaction | 3 months postoperative
  Determining patient specific factors by use of validated questionnaires
Patient Satisfaction | 6 months postoperative
  Determining patient specific factors by use of validated questionnaires
Patient Satisfaction | 1 year postoperative
  Determining patient specific factors by use of validated questionnaires
Patient Satisfaction | 2 years postoperative
  Determining patient specific factors by use of validated questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, Belgium